CLINICAL TRIAL: NCT07127679
Title: The Effect of Breast Milk on Pain and Stress During Retinopathy of Prematurity Examination
Brief Title: The Effect of Breast Milk on Pain and Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Emel BULDUR, clinical nursing, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1462/1442
Record Dates: First submitted 2025-08-07; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Breastfeeding; Retinopaty of Prematurity; Pain; Stress
Keywords: Retinopathy of Prematurity; ROP; Breast Milk; Pain; Stress
MeSH Terms: conditions — Breast Feeding; Pain; Retinopathy of Prematurity | interventions — Pregnane X Receptor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- breast milk group (Experimental): Two minutes before the ROP examination, 2mL of freshly expressed breast milk was administered to infants in the experimental group using a syringe, placing the milk on the front of the tongue. As part of routine care, all infants were swaddled and given a pacifier before the procedure. Video recording began 3 minutes prior to the ROP examination and continued until the infant stopped crying post-examination.
  Interventions: Other: Two minutes before the ROP examination, 2 mL of freshly expressed breast milk was administered to infants in the experimental group using a syringe, placing the milk on the front of the tongue. As par
- control group (No Intervention): As part of routine care, all infants were swaddled and given a pacifier before the procedure. Video recording began 3 minutes prior to the ROP examination and continued until the infant stopped crying post-examination.

INTERVENTIONS:
Other: Two minutes before the ROP examination, 2 mL of freshly expressed breast milk was administered to infants in the experimental group using a syringe, placing the milk on the front of the tongue. As par — Data were collected using the premature infant information form, the premature infant vital signs record form, the Premature Infant Pain Profile (PIPP), and the Neonatal Stress Scale. Two minutes before the ROP examination, 2mL of freshly expressed breast milk was administered to infants in the experimental group using a syringe, placing the milk on the front of the tongue. As part of routine care, all infants were swaddled and given a pacifier before the procedure. Video recording began 3 minutes prior to the ROP examination and continued until the infant stopped crying post-examination. Recordings were assessed by two independent observers to determine pain and stress scores, as well as parameters such as heart rate, oxygen saturation, perfusion index, and duration of crying.
  Arms: breast milk group

SUMMARY:
This study aimed to examine the effect of breast milk on pain and stress during Retinopathy of Prematurity (ROP) examinations. This randomized controlled experimental study was conducted with premature infants (N = 154) hospitalized in the Department of Child Health and Diseases, Neonatology Unit, at Izmir Ege University Faculty of Medicine Hospital between February 2024 and January 2025. A total of 36 premature infants (experimental group: 18; control group: 18) who met the inclusion criteria were included in the study. Data were collected using the Infant Information Form, the Premature Infant Pain Profile (PIPP), and the Neonatal Stress Scale. Two minutes before the ROP examination, 2 mL of freshly expressed breast milk was administered to infants in the experimental group using a syringe, placing the milk on the front of the tongue. Breast milk may be effective in reducing pain and stress associated with ROP examinations.

Keywords: Retinopathy of Prematurity; ROP; Breast Milk; Pain; Stress

DETAILED DESCRIPTION:
This study aimed to examine the effect of breast milk on pain and stress during Retinopathy of Prematurity (ROP) examinations. This randomized controlled experimental study was conducted with premature infants (N = 154) hospitalized in the Department of Child Health and Diseases, Neonatology Unit, at Izmir Ege University Faculty of Medicine Hospital between February 2024 and January 2025. A total of 36 premature infants (experimental group: 18; control group: 18) who met the inclusion criteria were included in the study. Data were collected using the premature infant information form, the premature infant vital signs record form, the Premature Infant Pain Profile (PIPP), and the Neonatal Stress Scale. Two minutes before the ROP examination, 2 mL of freshly expressed breast milk was administered to infants in the experimental group using a syringe, placing the milk on the front of the tongue. As part of routine care, all infants were swaddled and given a pacifier before the procedure. Video recording began 3 minutes prior to the ROP examination and continued until the infant stopped crying post-examination. Recordings were assessed by two independent observers to determine pain and stress scores, as well as parameters such as heart rate, oxygen saturation, perfusion index, and duration of crying.

The study found that pain scores were significantly lower in the group that received breast milk prior to the ROP examination compared to the control group (p <0.001). Stress scores were also significantly lower in the breast milk group (p < 0.001).The breast milk group showed more favorable oxygen saturation and heart rate levels (p < 0.05). There was no significant difference in perfusion index between the two groups. Crying duration was significantly shorter in the breast milk group compared to the control group (p < 0.001). Breast milk may be effective in reducing pain and stress associated with Retinopathy of Prematurity examinations.

ELIGIBILITY:
Inclusion Criteria:

* The baby's birth week is ≤34 or birth weight is ≤1700 grams, room babies who are monitored in good mood and have good clinical findings
* Babies who have developed sucking and swallowing skills and can hold a pacifier
* Any analgesic, muscle relaxant and sedative that may affect the pain level not taking effective medication
* The family agrees to participate in the study.
* Babies are in neonatal intensive care
* Having babies who are exclusively breastfed
* First ROP examination

Exclusion Criteria:

* Babies with congenital anomalies and metabolic diseases, cleft palate and cleft babies with lips did not sign the informed consent form and did not participate in the study.
* Babies from families that did not accept were not included in the study.

Ages: 30 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Premature Infant Pain Profile (PIPP), | one week
  The Premature Infant Pain Profile (PIPP) is a behavioral measure of pain for premature infants. It was developed at the Universities of Toronto and McGill in Canada. Minimum score: 0, maximum score: 21.The higher the score the greater the pain behavior.The PIPP is a 7-item multidimensional (composite) measure of pain that has been used widely to assess acute pain in infants. The PIPP includes 3 behavioral (facial actions: brow bulge, eye squeeze, nasolabial furrow), 2 physiological (heart rate and oxygen saturation), and 2 contextual (gestational age [GA] and behavioral state [BS]) items.
Neonatal Stress Scale | one week
  This scale is used in premature babies. It was prepared to evaluate stress. 8 subgroups (facial expression, body color, breathing, activity level, consolability, muscle tone, extremities, posture). The form consisting of 24 items is a 3-point Likert type. In the preparation of the draft form, the principles included in the Synactive Theory created within the framework of concepts.
  Each subgroup is scored between 0 and 2. The maximum score on the scale is 16, and the minimum is 0. A score of 0 indicates that the baby is not stressed. The higher the score, the higher the baby's stress level.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege Unversity, Bornova, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided